CLINICAL TRIAL: NCT03431324
Title: Employing Episodic Future Thinking About Mating Opportunities to Induce Lower Cigarette Consumption
Brief Title: Mating-EFT Smoking Cessation Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Dr. Michael Baker, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 18-0509
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Smoking Cessation; Motivation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Stage 1 will employ a between-subjects experimental design to establish the effectiveness of the mating-EFT intervention and compare its effectiveness to that of the established general-EFT intervention (Chiou & Wu, 2017) and a yoked control condition. This study will determine whether the effectiveness of these interventions is moderated by individual differences in relationship status, fundamental social motives (including mate-seeking motivation), self-efficacy, and nicotine dependence.
  Stage 2 will employ a quasi-experimental design in which participants who are either currently involved in a committed romantic relationship or single will be randomly assigned to complete either a mating-centric EFT intervention, a general-EFT intervention, or a control activity that involves no intervention.
Who Masked: Participant
Masking Description: Participants will be blind to the hypothesis of the study and to the condition to which they are assigned. They will be informed of both of these details during a debriefing provided by the researcher upon the conclusion of data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mating-EFT Intervention Effectiveness (Experimental): Study 1: 90 participants will attend an initial session, at which point they will provide demographic information as well as their relationship status. They will then be randomly assigned to complete either the Episodic Future Thinking about Mating Opportunities intervention, a general-EFT intervention, or an unrelated questionnaire (yoked control condition).
  All participants will submit daily reports of the number of cigarettes smoked for a period of one week. Participants will then complete a series of questionnaires measuring individual differences in fundamental social motives (including mate-seeking motives), self-efficacy, and nicotine dependence.
  Interventions: Behavioral: Episodic Future Thinking about Mating Opportunities
- Message Tailoring for Smoking Cessation (Experimental): Study 2: A quasi-experimental design will be employed in order to determine whether targeting individuals who are single and highly motivated to seek a mate with a Targeted Mating-EFT Intervention is a more effective means of reducing cigarette consumption than presenting all individuals with a general-EFT intervention. A total of 180 smokers who intend to quit or reduce smoking will be recruited as participants. These individuals will be selected from a larger pool of participants based upon responses to screening questions. The screening questions will measure relationship status and mate seeking motivation.
  Interventions: Behavioral: Targeted Mating-EFT Intervention

INTERVENTIONS:
Behavioral: Episodic Future Thinking about Mating Opportunities — Participants who complete the mating-EFT intervention will be instructed to write about three positive mating-related events that would occur within the course of one year "if you successfully quit smoking now." Participants will then be asked to close their eyes and imagine the events that they listed as specifically and vividly as possible (e.g., to imagine the setting and the sequence of the events, as well as the persons and objects that would be present. A period of one minute will be allotted for participants to mentally pre-experience each event.
  The general-EFT intervention will be structured similarly to, with the key exception of being instructed to write about and imagine three "positive life events".
  Arms: Mating-EFT Intervention Effectiveness
Behavioral: Targeted Mating-EFT Intervention — This intervention is identical to the "Episodic Future Thinking about Mating Opportunities" intervention with the exception that in Arm 2 the aim will be to determine whether the Mating-EFT intervention is especially effective when administered to individuals who are single or highly motivated to seek a mate.
  Arms: Message Tailoring for Smoking Cessation

SUMMARY:
The current proposal aims to develop and establish the effectiveness of a novel behavioral smoking cessation intervention. Previous research has shown that having smokers engage in episodic future thinking (EFT) about specific positive life outcomes that they could experience if they quit smoking immediately can be an effective means of reducing cigarette consumption. This intervention allowed participants to generate their own general positive life outcomes. While the existing intervention approaches motivation from a generalist perspective, the current proposal seeks to modify this intervention to fit within a Fundamental Social Motives (FSM) framework. The FSM framework posits that there exist individual differences in fundamental social motives such as self-protection, disease avoidance, affiliation, kin care, and mating motives such that some individuals are more motivated to work toward some of these goals than others. Specifically, the current proposal seeks to develop an EFT intervention that appeals to fundamental mating motives by asking participants to imagine positive mating outcomes that they might experience in one year's time if they were to quit smoking immediately. This will be accomplished via two empirical studies. Study 1 will compare the effectiveness of the mating-EFT intervention to the general-EFT intervention and a yoked control condition while examining the possibility that individual differences in relationship status, mating motives, self-efficacy, and nicotine dependence moderate these effects. Study 2 will employ a quasi-experimental design to test the effectiveness of this intervention using a tailored messaging approach, assigning smokers who are either single and motivated to seek new mates or involved in a committed relationship and not motivated to seek new mates to complete the general or mating-EFT or a control task. The investigators predict that the mating-EFT will be more effective than the general EFT in reducing cigarette consumption, particularly if it is administered to participants who have more active mating goals.

DETAILED DESCRIPTION:
Tobacco use is one of the leading causes of preventable illness and premature death worldwide. Individuals who smoke tobacco tend to develop a physical addiction to nicotine. Behavioral interventions have been shown to be an effective means of assisting with smoking cessation. Smoking cessation interventions, especially those of a brief and intensive nature, have been shown to be a cost-effective means of preventing negative health outcomes and extending life expectancy.

The PRIME theory of motivation regards cigarette addiction as a disorder of motivation. Accordingly, this theory seeks to help practitioners to identify effective means of overcoming addition through an analysis of the plans, responses, motives, impulses, and evaluations of smokers. Behavioral interventions often employ motivation interviewing with the goal of enhancing the motivation of smokers to quit by increasing their enthusiasm for positive life outcomes associated with quitting as well as giving a sense of purpose to this behavioral change.

Evolutionary perspectives on human behavior suggest that the desire to find a mate is a fundamental social motive that drives much of human behavior. Accordingly, encouraging smokers to think about how quitting could be beneficial to their mating goals could be an effective means of enhancing motivation to quit. A brief intervention that requires smokers to employ episodic future thinking (EFT) has been shown to effectively reduce smoking behavior. The current proposal aims to (1) develop and test the effectiveness of a behavioral intervention that employs EFT about how immediate quitting of smoking could enhance prospects for mating success and (2) refine this intervention by identifying key individual differences that impact its effectiveness, in order to maximize successful cessation outcomes by targeting populations that would be more strongly motivated by mating-related goals.

Aim 1: To develop and test the effectiveness of a behavioral smoking cessation intervention that employs EFT about future mating opportunities. EFT involves thinking about oneself experiencing a specific future event. Research indicates that this type of thinking reduces the tendency for people to discount the future costs associated with current behaviors and to reduce cigarette consumption. Since mating goals are of fundamental importance to human social life, an intervention that involves EFT about how quitting smoking could lead to increased likelihood of success in a specific future mating situation may be an especially effective means of motivating smokers to quit. Specifically, smokers will be instructed to imagine how quitting today could improve their chances of attracting a mate in a specific future mating situation.

Aim 2: To determine whether individual differences in mating motives moderate the effectiveness of the proposed intervention. People who are involved in a committed romantic relationship are often less motivated to seek a new mate than people who are single. Furthermore, some people are generally more motivated to seek new mates than others, regardless of relationship status. Self-report measures are commonly used to measure individual differences in preference for sexual variety and motivation to seek new mates. The investigators aim to determine whether relationship status and mating motivation moderate the effectiveness of the proposed mating-EFT smoking cessation intervention. The investigators predict that this intervention would be most effective among individuals who are not currently involved in a committed romantic relationship and are highly motivated to seek new mates.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Fluent in English
* Current smoker

  * Motivated to quit or reduce their cigarette consumption

Exclusion Criteria:

* Under 18 years of age
* Not fluent in English
* Not currently a smoker

  * Not motivated to quit or reduce cigarette consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Cigarette Consumption | 7 days
  During the initial session, participants will be asked to report how many cigarettes they smoke during a typical week. This will serve as a baseline to which the number of cigarettes smoked following exposure to the interventions will be compared. This within-subjects comparison will complement the between-subjects comparison that will be used in order to test the effectiveness of the manipulation within each group.

SECONDARY OUTCOMES:
Motivation to Quit or Reduce Smoking | 7 days
  Participants will also report their level of motivation to quit smoking or reduce their cigarette consumption as well as how motivated they are by different positive life outcomes that could result from quitting. This measurement will serve as both a manipulation check (with participants in the mating-EFT condition expected to report that they are more motivated by mating-related benefits of smoking cessation compared to the other conditions) as well as a secondary dependent variable that will also allow us to determine whether motivation is a mechanism influencing smoking cessation efforts.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Baker, Ph.D., Principal Investigator — East Carolina University

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized IPD may be shared with other researchers following publication of the results of this work. A sequentially generated code number will be provided to participants that will be used during data collection in lieu of their name in the interest of protecting participant privacy. This code number will be included in any shared data.

REFERENCES:
- [Background] Chiou WB, Wu WH. Episodic Future Thinking Involving the Nonsmoking Self Can Induce Lower Discounting and Cigarette Consumption. J Stud Alcohol Drugs. 2017 Jan;78(1):106-112. doi: 10.15288/jsad.2017.78.106. PMID 27936370